CLINICAL TRIAL: NCT01135095
Title: Validation of a Low-Dose One-Day TC99m Protocol With a High-Efficiency Cardiac Dedicated Gamma Camera for Detection of Coronary Artery Disease
Brief Title: Low Dose One-Day Tc99m Protocol With a High-Efficiency Cardiac Dedicated Gamma Camera For Detection of Coronary Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Spectrum Dynamics (Industry)
Collaborators: PeaceHealth Medical Group (Other); Brigham and Women's Hospital (Other); Cedars-Sinai Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SD-DSPECT002
Record Dates: First submitted 2009-10-15; First posted 2010-06-02 (Estimated); Results first posted 2021-01-26 (Actual); Last update posted 2021-01-26 (Actual); Status verified 2021-01

CONDITIONS: Chest Pain
Keywords: Myocardial perfusion; Low radiation dose; Single photon emission computed tomography
MeSH Terms: conditions — Chest Pain | interventions — X-Rays

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- low-dose imaging (Experimental): low dose versus standard dose imaging
  Interventions: Radiation: low-dose imaging

INTERVENTIONS:
Radiation: low-dose imaging — The study is designed to assess the validity of a low dose (~5mSv) Tc99m one day protocol using D-SPECT standard protocol as the comparators.
  D-SPECT cardiac scanner the D-SPECT system uses a solid-state detector, made of an alloy of Cadmium, Zinc, and Telluride, eliminating the need for thick crystals and large photomultiplier tubes. As a result, the system is significantly miniaturized, and ergonomically optimized to both user and patient
  Other Names: low dose imaging

SUMMARY:
A prospective single clinical trial to validate the use of a low-dose (~5mSv) Tc-99m protocol with a high-efficiency cardiac dedicated camera (Dynamic Single Photon Emission Computed Tomography; D-SPECT) to detect myocardial perfusion abnormalities during myocardial perfusion imaging.

DETAILED DESCRIPTION:
as above

ELIGIBILITY:
Inclusion Criteria:

1. Patient is referred to myocardial perfusion D-SPECT for clinical indications.
2. Written informed consent is obtained by a study investigator.

Exclusion Criteria:

1. Patient is diagnosed as having uncontrolled congestive cardiac failure or cardiogenic shock.
2. Patient is diagnosed as having uncontrolled hypertension with resting blood pressure > 220 mm Hg systolic or 110 mm Hg diastolic.
3. Patient pregnancy (known or suspected).
4. Lack of written informed consent
5. Prisoner status
6. Minors under the age of 18 as coronary artery disease is generally an adult disease

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2010-06; Primary Completion 2012-06 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Einstein, MD,PHD, Principal Investigator — Columbia University Medical Center, Department of Medicine, Division of Cardiology; Dan Berman, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (2):
- United States (2):
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Oregon Heart and Vascular Institute, Springfield, Oregon

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 101 patients prospectively enrolled at 3 US hospital sites (Cedars-Sinai Medical Center, Oregon Heart and Vascular Institute, Brigham and Women's Hospital) between June 2010 and June 2012.
Pre-assignment Details: No post-enrollment pre-assignment significant events occurred.
Groups:
- Low-dose Imaging: Low-dose versus standard-dose imaging
  Low-dose imaging: the study is designed to assess the validity of a low-dose (~5mSv) Tc99m one day protocol using D-SPECT standard protocol as the comparators.
  D-SPECT cardiac scanner: the D-SPECT system uses a solid-state detector, made of an alloy of Cadmium, Zinc, and Telluride, eliminating the need for thick crystals and large photomultiplier tubes. As a result, the system is significantly miniaturized, and ergonomically optimized to both user and patient.
Period: Overall Study
Arm/Group | Low-dose Imaging
Started | 101
Completed | 101
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Patients with suspected or known coronary artery disease scheduled to undergo rest-stress 1 day 99mTc-based SPECT myocardial perfusion imaging.
Groups:
- Low-dose Imaging: Low-dose versus standard dose imaging
  Low-dose imaging: the study is designed to assess the validity of a low dose (~5mSv) Tc99m one day protocol using D-SPECT standard protocol as the comparators.
  D-SPECT cardiac scanner: the D-SPECT system uses a solid-state detector, made of an alloy of Cadmium, Zinc, and Telluride, eliminating the need for thick crystals and large photomultiplier tubes. As a result, the system is significantly miniaturized, and ergonomically optimized to both user and patient.
Arm/Group | Low-dose Imaging
Number analyzed (Participants) | 101
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.8 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47
  Male | 54
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 101
BMI [Mean (Standard Deviation); unit: Kg/m^2] | 26.1 (2.8)
Diabetes Mellitus [Count of Participants; unit: Participants] | 26
Hypertension [Count of Participants; unit: Participants] | 74
Hyperlipidemia [Count of Participants; unit: Participants] | 77
Current smoker [Count of Participants; unit: Participants] | 13
Family history of premature heart disease [Count of Participants; unit: Participants] | 31

OUTCOME MEASURES:

1. Primary Outcome: Summed Rest Score (SRS) Using American Heart Association 17 Segment Polar Map Model
Description: SRS is used to quantify presence/severity of SPECT rest myocardial perfusion defects, as assessed by visual analysis using American Heart Association (AHA) 17 segment polar map model; each segment correlates to a myocardial location. Perfusion abnormalities can be determined in relation to myocardial segment/s affected by ischemia and the perfusion defect severity scored using 0 - 4 scale for each segment (0, normal uptake; 1, mildly reduced uptake; 2, moderately reduced uptake; 3, severely reduced uptake; and 4, no uptake). SRS is calculated by summing individual scores from each of 17 segments to give an overall score between 0 and 68; a score of 0 indicates normal outcome and scores > 0 indicate increasingly worse outcomes as the score increases. For each patient, SRS will be compared between standard-low-dose (SLD) imaging from a conventional A-SPECT camera and ultra-low-dose (ULD) imaging from a high-efficiency D-SPECT camera, both acquired on the same day.
Time Frame: 1 day
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Low-dose Imaging
Number analyzed (Participants) | 101
score on a scale
  Summed Rest Score Ultra-Low-Dose High-Efficiency SPECT imaging: D-SPECT camera | 2.75 (5.41)
  Summed Rest Score Standard-Low-Dose A-SPECT imaging: Siemens ECAM/Symbia T6 or Philips Forte camera | 2.95 (5.40)

ADVERSE EVENTS:
Arm/Group | Low-dose Imaging
Serious Adverse Events (participants affected / at risk) | 0/101
Other Adverse Events (participants affected / at risk) | 0/101

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No